CLINICAL TRIAL: NCT01204671
Title: Partially-blind Immunogenicity and Safety Study of GSK Biologicals' Seasonal Influenza Vaccine GSK2321138A in Adults.
Brief Title: Safety and Immunogenicity Study of GSK Biologicals' Seasonal Influenza Candidate Vaccine (GSK2321138A)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114269
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2017-02

CONDITIONS: Influenza
Keywords: influenza infection; GSK Biologicals influenza vaccine GSK2321138A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- GSK2321138A Lot 1 Group (Experimental): Subjects received one dose of the GSK2321138A vaccine, Lot 1, at Day 0. The GSK2321138A vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza vaccine GSK2321138A
- GSK2321138A Lot 2 Group (Experimental): Subjects received one dose of the GSK2321138A vaccine, Lot 2, at Day 0. The GSK2321138A vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza vaccine GSK2321138A
- GSK2321138A Lot 3 Group (Experimental): Subjects received one dose of the GSK2321138A vaccine, Lot 3, at Day 0. The GSK2321138A vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza vaccine GSK2321138A
- Fluarix Group (Active Comparator): Subjects received one dose of the Fluarix™ vaccine at Day 0. The Fluarix™ vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: FluarixTM
- GSK2604409A Group (Active Comparator): Subjects received one dose of the GSK2604409A vaccine at Day 0. The GSK2604409A vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza vaccine GSK2604409A

INTERVENTIONS:
Biological: Influenza vaccine GSK2321138A — One intramuscular injection
  Arms: GSK2321138A Lot 1 Group; GSK2321138A Lot 2 Group; GSK2321138A Lot 3 Group
Biological: FluarixTM — One intramuscular injection
  Arms: Fluarix Group
Biological: Influenza vaccine GSK2604409A — One intramuscular injection
  Arms: GSK2604409A Group

SUMMARY:
This study is designed to assess the safety and immunogenicity of a GSK Biologicals' investigational vaccine GSK2321138A in adults 18 years old and older. This study is also designed to assess the lot-to-lot consistency of vaccine GSK2321138A. The blinding will be double blind for all groups except for the GSK2604409A Group which will be open.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 years of age or older at the time of the first vaccination
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Healthy subjects or those with chronic well-controlled disease as established by physical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* - has practiced adequate contraception for 30 days prior to vaccination,
* - and has a negative urine pregnancy test on the day of vaccination,
* and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of the study vaccine or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Administration of an influenza vaccine during the 6 months preceding entry into the study.
* Planned administration / administration of a vaccine not foreseen by the study protocol within 30 days before vaccination and up to Day 21.
* Any contra-indication to intramuscular administration of the influenza vaccines.
* History of hypersensitivity/anaphylaxis to a previous dose of influenza vaccine, history of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Any administration of a long-acting immune-modifying drug within 3 months before study start, or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease and/or fever at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* History of Guillain-Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* History of chronic alcohol consumption and/or drug abuse.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4659 (Actual)
Dates: Start 2010-10-04; Primary Completion 2011-06-06 (Actual); Study Completion 2011-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (10):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
- Germany (9):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Finsterwalde, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Berlin
- Romania (6):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Pantelimon
  - GSK Investigational Site, Ploieşti
- South Korea (4):
  - GSK Investigational Site, Guro Gu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (5):
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Vic/ Barcelona
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kieninger D, Sheldon E, Lin WY, Yu CJ, Bayas JM, Gabor JJ, Esen M, Fernandez Roure JL, Narejos Perez S, Alvarez Sanchez C, Feng Y, Claeys C, Peeters M, Innis BL, Jain V. Immunogenicity, reactogenicity and safety of an inactivated quadrivalent influenza vaccine candidate versus inactivated trivalent influenza vaccine: a phase III, randomized trial in adults aged >/=18 years. BMC Infect Dis. 2013 Jul 24;13:343. doi: 10.1186/1471-2334-13-343. PMID 23883186
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4659 subjects (all aged 18 years and older at the time of their first vaccination as part of this study) were enrolled in this study, of which 4656 were vaccinated. The study vaccine dose was not administrated but subject number was allocated for the other 3 subjects.
Pre-assignment Details: Subjects receiving the GSK2321138A and Fluarix™ vaccines were followed in a double-blinded manner throughout the entire study period, from Day 0 to Day 180. Subjects receiving the GSK2604409A vaccine were followed in an open manner until Day 21 only.
Period: Overall Study
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Started | 1012 | 1013 | 1011 | 1010 | 610
Completed | 998 | 998 | 998 | 997 | 606
Not Completed | 14 | 15 | 13 | 13 | 4
Not completed — Adverse Event | 4 | 3 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 5 | 3
Not completed — Lost to Follow-up | 7 | 8 | 6 | 4 | 0
Not completed — Unknown Completion Status | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group | Total
Number analyzed (Participants) | 1012 | 1013 | 1011 | 1010 | 610 | 4656
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (17.90) | 58.0 (17.41) | 57.9 (17.80) | 58.1 (17.83) | 58.1 (17.92) | 58.0 (17.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 598 | 578 | 569 | 548 | 343 | 2636
  Male | 414 | 435 | 442 | 462 | 267 | 2020

OUTCOME MEASURES:

1. Primary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. HI antibodies assessed were antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria), and B/Brisbane/3/2007 (Yamagata) flu strains. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: At Day 0 (D 0), and at Day 21 (D 21)
Population: The analysis was performed on the According-to-Protocol cohort for Immunogenicity, which included all vaccinated and eligible subjects for whom data concerning immunogenicity outcome measures were available, and for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- GSK2321138A Group: Subjects received one dose of the GSK2321138A vaccine, Lot 1, 2 or 3, at Day 0. The GSK2321138A vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1809 | 608 | 534
Titer
  H1N1 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H1N1 Strain - D 0 | 14.7 [13.8 to 15.6] | 15.6 [14.1 to 17.3] | 14.4 [12.9 to 16.0]
  H1N1 Strain - D 21 | 201.1 [188.1 to 215.1] | 218.4 [194.2 to 245.6] | 213.0 [187.6 to 241.9]
  H3N2 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H3N2 Strain - D 0 | 34.0 [31.8 to 36.3] | 38.1 [34.1 to 42.7] | 35.7 [31.6 to 40.3]
  H3N2 Strain - D 21 | 314.7 [296.8 to 333.6] | 298.2 [268.4 to 331.3] | 340.4 [304.3 to 380.9]
  Victoria Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Victoria Strain - D 0 | 73.8 [69.1 to 78.8] | 73.6 [65.5 to 82.8] | 71.7 [63.4 to 81.0]
  Victoria Strain - D 21 | 404.6 [386.6 to 423.4] | 393.8 [362.7 to 427.6] | 258.5 [234.6 to 284.8]
  Yamagata Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Yamagata Strain - D 0 | 101.4 [94.5 to 108.8] | 100.9 [89.3 to 113.9] | 99.8 [87.7 to 113.5]
  Yamagata Strain - D 21 | 601.8 [573.3 to 631.6] | 386.6 [351.5 to 425.3] | 582.5 [534.6 to 634.7]

2. Primary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease
Description: A seroconverted subject was a vaccinated subject who had either a pre-vaccination hemagglutination inhibition (HI) antibody titer < 1:10 and a post-vaccination titer above or equal (>=) 1:40, or a pre-vaccination HI antibody titer >= 1:10 and at least a 4-fold increase in post-vaccination HI antibody titer. Antibodies assessed were HI antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria), and B/Brisbane/3/2007 (Yamagata) flu strains. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: At Day 21 (D 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1801 | 605 | 530
Participants
  H1N1 Strain - D 21 | 1396 | 467 | 425
  H3N2 Strain - D 21 | 1287 | 398 | 371
  Victoria Strain - D 21 | 1046 | 335 | 252
  Yamagata Strain - D 21 | 1112 | 276 | 313

3. Secondary Outcome: Number of Seropositive Subjects Against 4 Strains of Influenza Disease
Description: A seropositive subject was a vaccinated subject with hemagglutination inhibition (HI) antibody titer above or equal (>=) the reference cut-off value of 1:10. Antibodies assessed were HI antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria), and B/Brisbane/3/2007 (Yamagata) flu strains. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: At Day 0 (D 0), and at Day 21 (D 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1809 | 608 | 534
Participants
  H1N1 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H1N1 Strain - D 0 | 967 | 352 | 291
  H1N1 Strain - D 21 | 1738 | 586 | 514
  H3N2 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H3N2 Strain - D 0 | 1416 | 488 | 425
  H3N2 Strain - D 21 | 1783 | 594 | 528
  Victoria Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Victoria Strain - D 0 | 1541 | 511 | 452
  Victoria Strain - D 21 | 1795 | 601 | 518
  Yamagata Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Yamagata Strain - D 0 | 1554 | 525 | 457
  Yamagata Strain - D 21 | 1794 | 597 | 532

4. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease
Description: A seroprotected subject was a vaccinated subject who had hemagglutination inhibition (HI) antibody titer above or equal (>=) 1:40. Antibodies assessed were HI antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria), and B/Brisbane/3/2007 (Yamagata) flu strains. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: At Day 0 (D 0), and at Day 21 (D 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1809 | 608 | 534
Participants
  H1N1 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H1N1 Strain - D 0 | 514 | 167 | 139
  H1N1 Strain - D 21 | 1651 | 558 | 495
  H3N2 Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  H3N2 Strain - D 0 | 965 | 353 | 285
  H3N2 Strain - D 21 | 1751 | 583 | 517
  Victoria Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Victoria Strain - D 0 | 1423 | 477 | 412
  Victoria Strain - D 21 | 1788 | 599 | 513
  Yamagata Strain - D 0: number analyzed (Participants) | 1801 | 605 | 530
  Yamagata Strain - D 0 | 1494 | 497 | 441
  Yamagata Strain - D 21 | 1792 | 595 | 532

5. Secondary Outcome: Increase in Hemagglutination Inhibition Antibodies Against 4 Strains of Influenza Disease
Description: Increase in hemagglutination inhibition (HI) antibodies is presented in terms of mean geometric increase (MGI), defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer , expressed using "fold increase" as unit . Antibodies assessed were HI antibodies against the A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2), B/Brisbane/60/2008 (Victoria), and B/Brisbane/3/2007 (Yamagata) flu strains. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: At Day 21 (D 21)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1801 | 605 | 530
fold change
  H1N1 Strain - D 21 | 13.69 [12.70 to 14.76] | 13.92 [12.23 to 15.84] | 14.88 [12.91 to 17.16]
  H3N2 Strain - D 21 | 9.28 [8.64 to 9.96] | 7.84 [6.93 to 8.88] | 9.52 [8.33 to 10.89]
  Victoria Strain - D 21 | 5.48 [5.12 to 5.85] | 5.37 [4.75 to 6.06] | 3.60 [3.25 to 3.98]
  Yamagata Strain - D 21 | 5.93 [5.53 to 6.36] | 3.84 [3.42 to 4.30] | 5.84 [5.13 to 6.65]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms post vaccination were pain, redness and swelling at the injection site. Any = occurrence of a symptom regardless of intensity. Grade 3 pain = significant pain at rest/ that prevented normal every day activities. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects, solely on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1008 | 1003 | 1004 | 1003 | 607
Participants
  Any Pain | 377 | 362 | 357 | 369 | 190
  Grade 3 Pain | 13 | 6 | 5 | 12 | 3
  Any Redness | 24 | 12 | 22 | 17 | 12
  Grade 3 Redness (≥ 100 mm) | 0 | 1 | 0 | 0 | 0
  Any Swelling | 26 | 20 | 16 | 21 | 8
  Grade 3 Swelling (≥ 100 mm) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: Assessed solicited local symptoms post vaccination were pain, redness and swelling at the injection site.
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 377 | 362 | 357 | 369 | 190
Day
  Pain | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Redness: number analyzed (Participants) | 24 | 12 | 22 | 17 | 12
  Redness | 2.0 [1.0 to 2.5] | 2.5 [1.5 to 4.5] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.5]
  Swelling: number analyzed (Participants) | 26 | 20 | 16 | 21 | 8
  Swelling | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.5 to 3.0] | 2.0 [1.0 to 3.0] | 2.5 [1.0 to 3.0]

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms post vaccination were fatigue, gastrointestinal symptoms (Gastr.), headache, joint pain at other location (Joint Pain), muscle aches, shivering, and temperature [axillary temperature above or equal to (>=) 37.5 degrees Celsius (°C)]. Any = occurrence of a symptom regardless of intensity or relationship to vaccination. Grade 3 = symptom which prevented normal every day activities. Grade 3 temperature = axillary temperature > 39°C. Related = symptom assessed as causally related to study vaccination.
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1008 | 1001 | 1002 | 1003 | 607
Participants
  Any Fatigue | 152 | 154 | 171 | 185 | 90
  Grade 3 Fatigue | 9 | 4 | 8 | 6 | 3
  Related Fatigue | 109 | 107 | 118 | 132 | 64
  Any Gastr. | 64 | 63 | 70 | 65 | 36
  Grade 3 Gastr. | 5 | 3 | 3 | 2 | 2
  Related Gastr. | 37 | 34 | 38 | 35 | 19
  Any Headache | 163 | 162 | 155 | 164 | 80
  Grade 3 Headache | 10 | 8 | 8 | 8 | 4
  Related Headache | 87 | 92 | 98 | 97 | 48
  Any Joint Pain | 96 | 84 | 74 | 104 | 57
  Grade 3 Joint Pain | 6 | 5 | 3 | 7 | 2
  Related Joint Pain | 67 | 54 | 51 | 61 | 29
  Any Muscle Aches | 165 | 172 | 156 | 195 | 98
  Grade 3 Muscle Aches | 5 | 2 | 7 | 8 | 3
  Related Muscle Aches | 117 | 130 | 109 | 137 | 61
  Any Shivering | 45 | 32 | 48 | 50 | 26
  Grade 3 Shivering | 3 | 2 | 6 | 3 | 1
  Related Shivering | 31 | 19 | 32 | 30 | 19
  Any Temperature (≥ 37.5°C) | 19 | 21 | 8 | 12 | 9
  Grade 3 Temperature (> 39.0°C) | 0 | 0 | 0 | 0 | 0
  Related Temperature | 11 | 16 | 3 | 5 | 6

9. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: Assessed solicited general symptoms post vaccination were fatigue, gastrointestinal symptoms (Gastr.), headache, joint pain at other location (Joint Pain), muscle aches, shivering, and temperature [defined as axillary temperature above or equal to (≥) 37.5 degrees Celsius (°C)].
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Day
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 165 | 172 | 171 | 195 | 98
Day
  Fatigue: number analyzed (Participants) | 152 | 154 | 171 | 185 | 90
  Fatigue | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Gastr.: number analyzed (Participants) | 64 | 63 | 70 | 65 | 36
  Gastr. | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.5]
  Headache: number analyzed (Participants) | 163 | 162 | 155 | 16 | 80
  Headache | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Joint Pain: number analyzed (Participants) | 96 | 84 | 74 | 104 | 57
  Joint Pain | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Muscle Aches | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Shivering: number analyzed (Participants) | 45 | 32 | 48 | 50 | 26
  Shivering | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Temperature: number analyzed (Participants) | 19 | 21 | 8 | 12 | 9
  Temperature | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs cover any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any unsolicited AE = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 unsolicited AE = unsolicited AE that prevented normal everyday activity Related unsolicited AE = unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 21-day (Days 0-20) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1012 | 1013 | 1011 | 1010 | 610
Participants
  Any Unsolicited AE(s) | 125 | 120 | 134 | 138 | 92
  Grade 3 Unsolicited AE(s) | 11 | 12 | 16 | 7 | 2
  Related Unsolicited AE(s) | 17 | 20 | 27 | 26 | 14

11. Secondary Outcome: Number of Subjects With Any and Related Adverse Events With Medically-attended Events (MAEs)
Description: Medically-attended events (MAEs) refer to non-serious and serious events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. If a MAE was leading to hospitalisation (or met any other serious adverse event criterion), it was reported as serious adverse event. Related MAE = MAE assessed by the investigator as related to the vaccination. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: From the beginning of the study (Day 0) to study end (Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Fluarix Group: Subjects received one dose of the Fluarix™ vaccine at Day 0. The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 3036 | 1010 | 610
Participants
  Any MAE(s) | 688 | 216 | 52
  Related MAE(s) | 11 | 4 | 5

12. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of adverse events that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Related pIMD = pIMD assessed by the investigator as related to the vaccination. Subjects receiving the GSK2321138A vaccine were pooled for this outcome measure.
Time Frame: From the beginning of the study (Day 0) to study end (Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 3036 | 1010 | 610
Participants
  Any pIMD(s) | 1 | 1 | 0
  Related pIMD(s) | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE = any SAE regardless of intensity or relationship to vaccination. Related SAE = SAE assessed by the investigator as related to the vaccination.
Time Frame: From the beginning of the study (Day 0) to study end (Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 1012 | 1013 | 1011 | 1010 | 610
Participants
  Any SAE(s) | 28 | 20 | 22 | 26 | 1
  Related SAE(s) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: Within the 7-day (Days 0-6) follow-up period after vaccination. Unsolicited adverse events: Within the 21-day (Days 0-20) follow-up period after vaccination. Serious adverse events: Throughout the study period (Days 0 to 180)
Description: Analysis for unsolicited AEs and SAEs was performed on all vaccinated subjects, and analysis for solicited symptoms was performed solely on vaccinated subjects for whom results were available.
Groups:
- Fluarix Group: Subjects received one dose of the 1 dose of the Fluarix™ vaccine at Day 0. The Fluarix™ vaccine was administered as a single dose intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2321138A Lot 1 Group | GSK2321138A Lot 2 Group | GSK2321138A Lot 3 Group | Fluarix Group | GSK2604409A Group
Serious Adverse Events (participants affected / at risk) | 28/1012 | 20/1013 | 22/1011 | 26/1010 | 1/610
Other Adverse Events (participants affected / at risk) | 485/1008 | 472/1003 | 482/1004 | 500/1003 | 275/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2321138A Lot 1 Group (N=1012) | GSK2321138A Lot 2 Group (N=1013) | GSK2321138A Lot 3 Group (N=1011) | Fluarix Group (N=1010) | GSK2604409A Group (N=610)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 2 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Central nervous system infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ammonia increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Rectal cancer ( (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 2 | 2 | 0
Coma hepatic (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2321138A Lot 1 Group (N=1008) | GSK2321138A Lot 2 Group (N=1003) | GSK2321138A Lot 3 Group (N=1004) | Fluarix Group (N=1003) | GSK2604409A Group (N=607)
Pain (General disorders) | 377 | 362 | 357 | 369 | 190
Fatigue (General disorders) | 152 | 154 | 171 | 185 | 90
Gastrointestinal symptoms (General disorders) | 64 | 63 | 70 | 65 | 36
Headache (General disorders) | 163 | 162 | 155 | 164 | 80
Joint pain (General disorders) | 96 | 84 | 74 | 104 | 57
Muscle aches (General disorders) | 165 | 172 | 156 | 195 | 98

LIMITATIONS AND CAVEATS:
Concerns arose about data integrity for a Romanian site (102 subjects) after completion of analysis. These data were not excluded from this reporting as they did not reveal irregularities and GSK does not plan to use them towards regulatory filing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.